CLINICAL TRIAL: NCT03128671
Title: Reorientation Intervention for Delirium in ICU
Brief Title: Family Automated Voice Reorientation Study
Acronym: FAVoR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: University of South Florida (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Cindy Munro, Dean and Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20170771; Pro00027039 (Other: USF IRB); R01NR016702 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-04-25 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Delirium; Cognitive Impairment; Health, Subjective; Sleep
Keywords: intensive care unit; critical care; mechanical ventilation; confusion; polysomnography; delirium; adult
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Confusion

STUDY DESIGN:
Intervention Model Description: prospective, randomized, experimental design
Who Masked: Outcomes Assessor
Masking Description: Study personnel evaluating delirium will use standardized tool (CAM-ICU) and will be blinded to subjects' group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAVoR Intervention Group (Experimental): In the intervention group, scripted audio messages recorded by the patient's family (FAVoR intervention) will be played for the patient at hourly intervals during daytime hours. These messages will be personalized, delivered automatically, and provide information about the ICU environment. The FAVoR intervention, a standardized protocol developed and tested in preliminary work, will be delivered by audio recording for 5 consecutive days (120 hours), or until ICU discharge if discharge occurs within the first 5 days. The number of episodes of delirium during ICU stay is the primary outcome measure. Data will also be collected at 1 month and 6 months following hospital discharge for secondary aim 3.
  Interventions: Behavioral: FAVoR Intervention
- Control Group (No Intervention): The control group will not receive the FAVoR intervention. The number of episodes of delirium during ICU stay is the primary outcome measure. Data will also be collected at 1 month and 6 months following hospital discharge for secondary aim 3.

INTERVENTIONS:
Behavioral: FAVoR Intervention — The FAVoR intervention includes a set of 8 scripted recorded messages, no longer than 2 minutes long, includes subject's name, uses simple terms, and is written at a 5th grade reading level. Messages include information about the critical care environment, the visual and auditory stimuli to be expected, and the availability of providers and family.
  Arms: FAVoR Intervention Group

SUMMARY:
This randomized clinical trial tests a cognitive reorientation intervention to prevent delirium in the intensive care unit using scripted audio messages, recorded by the patient's family and played at hourly intervals during daytime hours, to provide information about the ICU environment to the patient (the Family Automated Voice Reorientation intervention, FAVoR). The investigators hypothesize that providing ongoing orientation to the ICU environment through recorded audio messages in a voice familiar to the patient will enable the patient to more accurately interpret the environment and reduce risk of delirium. Increasing awareness of daytime by cuing patients during waking hours may also improve day/night orientation, nighttime sleep/rest, and further reduce risk of delirium.

DETAILED DESCRIPTION:
This randomized clinical trial will test the effectiveness of a nonpharmacologic intervention to prevent delirium in the intensive care unit (ICU), which affects as many as 80% of critically ill, mechanically ventilated adults.. The Family Automated Voice Reorientation (FAVoR) intervention uses scripted audio messages, recorded by the patient's family and played at hourly intervals during daytime hours, to provide information about the ICU environment to the patient; this ongoing orientation to the ICU environment through recorded messages in a voice familiar to the patient may enable the patient to more accurately interpret the environment and thus reduce risk of delirium. Increasing awareness of daytime by cuing patients during waking hours may also improve day/night orientation and nighttime sleep, further reducing risk of delirium. The primary specific aim of the project is to test the effect of the FAVoR intervention on delirium in critically ill, mechanically ventilated adults during hospitalization in the ICU. Secondary aims are to: (1) explore if the effect of FAVoR on delirium is mediated by sleep, (2) explore if selected biobehavioral factors may potentially moderate the effects of FAVoR on delirium, and (3) examine the effects of FAVoR on short term (immediately after ICU discharge) and long term (1 and 6 months after hospital discharge) outcomes, including cognitive function and patient-reported health status.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients
* within 36 hours of ICU admission
* patient or legally authorized representative (LAR) must be able to provide informed consent in English or Spanish
* a family member able to speak English or Spanish must be available and willing to audio record scripted messages

Exclusion Criteria:

* dementia (because it complicates planned longitudinal cognitive assessments)
* anticipation by the clinical provider of imminent patient death
* medical contraindication to the intervention (for example, psychiatric history of auditory hallucinations, or profoundly deaf)
* inability to speak either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Munro, PhD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - University of Miami UHealth Tower, Miami, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munro CL, Liang Z, Elias MN, Ji M, Chen X, Kip PL, Greengold J, Ely EW, Calero K. Delirium Reduction via Scripted Family Voice Recordings in Critically Ill Patients Receiving Mechanical Ventilation. Am J Crit Care. 2025 Nov 1;34(6):429-437. doi: 10.4037/ajcc2025486. PMID 41173649
- [Derived] Munro CL, Liang Z, Elias MN, Ji M, Chen X, Calero K. Sleep and Activity Patterns Are Altered During Early Critical Illness in Mechanically Ventilated Adults. Dimens Crit Care Nurs. 2021 Jan-Feb 01;40(1):29-35. doi: 10.1097/DCC.0000000000000455. PMID 33560633

RESULTS

PARTICIPANT FLOW:
Period: Enrollment
Arm/Group | FAVoR Intervention Group | Control Group
Started | 89 | 89
Completed | 89 | 89
Not Completed | 0 | 0
Period: Allocation
Arm/Group | FAVoR Intervention Group | Control Group
Started | 89 | 89
Completed | 80 | 89
Not Completed | 9 | 0
Not completed — ICU discharge prior to intervention initiation | 4 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Period: Intervention
Arm/Group | FAVoR Intervention Group | Control Group
Started | 80 | 89
Completed | 44 | 55
Not Completed | 36 | 34
Not completed — Withdrawal by Subject | 11 | 10
Not completed — Palliative/hospice care initiated | 9 | 10
Not completed — Death | 13 | 11
Not completed — Interrupted by hurricane | 1 | 0
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FAVoR Intervention Group | Control Group | Total
Number analyzed (Participants) | 89 | 89 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.96 (16.78) | 60.62 (17.45) | 59.29 (17.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 40 | 71
  Male | 58 | 49 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 56 | 107
  Not Hispanic or Latino | 38 | 33 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 15 | 37
  White | 66 | 73 | 139
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Delirium-free Days
Description: Delirium will be assessed by study personnel, blinded to the group assignment, using Confusion Assessment Method-Intensive Care Unit (CAM-ICU)
Time Frame: Up to 20 days in the intensive care unit (ICU)
Population: Delirium assessment were not conducted for all participants due to the following reasons: subject remained deeply sedated and so did not pass criteria for proceeding with the Confusion Assessment Method - Intensive Care Unit (CAM-ICU) assessment and/or subject was extubated prior to the scheduled delirium assessment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FAVoR Intervention Group | Control Group
Number analyzed (Participants) | 44 | 43
days | 8.4 (9.07) | 7.2 (5.8)

2. Secondary Outcome: Sleep
Description: Sleep Profiler polysomnography
Time Frame: Up to 5 days in the ICU
Reporting Status: Not Posted

3. Secondary Outcome: Cognitive Function
Description: NIH Cognitive Toolbox measures
Time Frame: At least 24 hours post ICU discharge, 1 month post hospital discharge, & 6 months post hospital discharge
Reporting Status: Not Posted

4. Secondary Outcome: Patient-reported Health Status
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scales
Time Frame: At least 24 hours post ICU discharge, 1 month post hospital discharge, & 6 months post hospital discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | FAVoR Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 14/89 | 11/89
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 1/89 | 0/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAVoR Intervention Group (N=89) | Control Group (N=89)
Blood Pressure Fluctuation (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03128671/Prot_SAP_000.pdf